CLINICAL TRIAL: NCT01434420
Title: Triple Negative Breast Cancer: Study of Molecular and Genetic Factors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: SA03/IPC 2010-003
Record Dates: First submitted 2011-09-13; First posted 2011-09-14 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-12

CONDITIONS: Breast Cancer
Keywords: triple negative breast cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Triple negative breast cancer (Experimental): Triple negative breast cancer
  Interventions: Genetic: BRCA1 BRCA2 PTEN PALB2 mutation

INTERVENTIONS:
Genetic: BRCA1 BRCA2 PTEN PALB2 mutation — detection of BRCA1 BRCA2 PTEN PALB2 mutation

SUMMARY:
Breast cancer triples negatives (TN; 15 % of the cases) are characterized by a high histoprognostic grade, a strong proliferation, a strong metastatic power, and a worse prognosis than the other forms of breast cancer. It is however a heterogenous group for histological and molecular level, but also for evolution. Most of the TN is part of the basal breast cancer subcategory. Until now, the medical treatment is based on chemotherapy.

Breast cancers by constitutional mutation of BRCA1 / BRCA2 (5 % of breast cancers) are mostly of basal type and their prognostic seems better that what could be expected from high grade tumours and without hormonal receptors. They would be much more frequent in the TN group. However, at this day, no prospective study was led to estimate this incidence, or to study the intervention of other genes of predisposition, as well to analyse the links between this phenotype and their consequences at the germinal or somatic level, in terms of associated molecular changes and prognosis.

The purpose of this study is, on a prospective study, to lead a joined analysis at the germinal level, in search of mutations of the main genes of breast cancer predisposition (BRCA1/2, PALB2, PTEN, PALB2), and at the tumour level (tissue micro-array and transcriptome), by correlating these results to the main clinical parameters.

The 5 years relapse-free survival will also be estimated.

ELIGIBILITY:
Inclusion Criteria:

* women > 18
* non metastatic breast cancer
* triple negative
* 5 years follow-up
* signed informed consent

Exclusion Criteria:

* other cancer (except in situ)
* metastases at diagnosis
* impossibility of follow-up

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-03; Primary Completion 2014-08 (Actual); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
incidence of BRCA1/2, PALB2, PTEN, PALB2 mutations | up to 1 month
  1) Determine the incidence of the BRCA1/2, PALB2, PTEN, PALB2 mutations in patients having at diagnosis a non metastatic triple negative breast cancer

SECONDARY OUTCOMES:
molecular profiles | up to 1 month
  2) Determine by tissue micro- array and transcriptome the molecular profiles and their correlation with the presence of a mutation
years relapse-free survival | at 5 years
  3) Determine the 5 years relapse-free survival in presence or not of a mutation, and according to the molecular profile of expression.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc EXTRA, MD, Principal Investigator — Institut Paoli-Calmettes
Locations (4):
- France (4):
  - Centre jean Perrin, Clermont-Ferrand
  - Hopital La Timone, Marseille
  - Institut Paoli-Calmettes, Marseille
  - Centre Antoine Lacassagne, Nice

REFERENCES:
- See also: sponsor web site — http://www.institutpaolicalmettes.fr/